CLINICAL TRIAL: NCT03364335
Title: A Randomized, Double-blind, Placebo-controlled Study of Effects of Two Fixed-dose Leucine-sildenafil Combinations (NS-0300) or Two Fixed-dose Leucine-sildenafil-metformin Combinations (NS-0200) Versus Placebo on Body Weight in Obesity
Brief Title: The Effect Of NS-0200 and NS-0300 Versus Placebo on Weight In Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NuSirt Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NS-WM-01
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Results first posted 2018-11-27 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2018-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double blind, placebo controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Each dose of placebo will consist of three tablets, identical in appearance to those used in the two active treatment arms, containing 93.5% Microcrystalline cellulose PH 102, 5.0% Crospovidone XL 10, 1.0% Silica gel (Syloid 244), 0.5% Magnesium stearate I MF3V for the leucine matched placebo and 99.5% Avicel PH200 , 0.5% magnesium stearate (w/w) and Opadry II White coating 3% weight gain for the sildenafil matched placebo.
  Interventions: Drug: Placebo
- Leu Sil 1.0mg (Experimental): 3 capsules BID consisting of 2 capsules containing 550 mg L-leucine each and 1 capsule containing 1.0 mg of sildenafil
  Interventions: Drug: Leu Sil 1.0mg; Drug: Leu Sil 4.0mg
- Leu Sil 4.0mg (Experimental): 3 capsules BID consisting of 2 capsules containing 550 mg L-leucine each and 1 capsule containing 4.0 mg of sildenafil
  Interventions: Drug: Leu Sil 1.0mg; Drug: Leu Met Sil 1.0mg
- Leu Met Sil 1.0mg (Experimental): 3 capsules BID consisting of 2 capsules containing 550 mg L-leucine and 250 mg metformin and 1 capsule containing 1.0 mg of sildenafil
  Interventions: Drug: Leu Sil 1.0mg; Drug: Leu Sil 4.0mg; Drug: Leu Met Sil 4.0mg
- Leu Met Sil 4.0mg (Experimental): 3 capsules BID consisting of 2 capsules containing 550 mg L-leucine and 250 mg metformin and 1 capsule containing 4.0 mg of sildenafil
  Interventions: Drug: Leu Sil 1.0mg; Drug: Leu Met Sil 1.0mg; Drug: Leu Met Sil 4.0mg

INTERVENTIONS:
Drug: Leu Sil 1.0mg — Leu 1100 mg + 1mg Sil BID
  Other Names: NS-0300-1.0
  Arms: Leu Met Sil 1.0mg; Leu Met Sil 4.0mg; Leu Sil 1.0mg; Leu Sil 4.0mg
Drug: Leu Sil 4.0mg — Leu 1100 mg + 4mg Sil BID
  Other Names: NS-0300-4.0
  Arms: Leu Met Sil 1.0mg; Leu Sil 1.0mg
Drug: Leu Met Sil 1.0mg — Leu 1100 mg + Met 500mg + 1mg Sil BID
  Other Names: NS-0200-1.0
  Arms: Leu Met Sil 4.0mg; Leu Sil 4.0mg
Drug: Leu Met Sil 4.0mg — Leu 1100 mg + Met 500mg + 4mg Sil BID
  Other Names: NS-0200-4.0
  Arms: Leu Met Sil 1.0mg; Leu Met Sil 4.0mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a 24-week study to evaluate the effects of two fixed-dose combinations of leucine and sildenafil or two fixed-dose combinations of leucine, sildenafil and metformin compared to placebo. The primary objective of this study is to evaluate the percentage change in body weight in subjects from Baseline/Visit 2 (Day 1) to Study Termination/Visit 8 (Day 168/Week 24).

DETAILED DESCRIPTION:
This is a randomized, 24-week, placebo-controlled, double-blind study to evaluate the effects of two fixed-dose combinations of leucine and sildenafil or two fixed-dose combinations of leucine, sildenafil and metformin compared to placebo. Subjects meeting all the inclusion criteria and no exclusion criteria will be randomized to one of five study arms.

The primary objective of this study is to evaluate the percentage change in body weight in subjects from Baseline/Visit 2 (Day 1) to Study Termination/Visit 8 (Day 168/Week 24) receiving two fixed-dose combinations of leucine and sildenafil or two fixed-dose combinations of leucine, sildenafil and metformin compared to placebo. Secondary objectives will also assess changes in absolute body weight, percentage of patients with ≥5% body weight loss, change in waist circumference, change in HbA1c, change in fasting glucose, change in blood lipids such as cholesterol, LDL, HDL, triglycerides, change in blood pressure and changes in in C-reactive protein. In addition this study will evaluate the safety and tolerability of NS-0200 and NS-0300.

Patients will have one screening visits which will determine their eligibility based on lab tests. Once qualified, patients will be randomly assigned to either one of the treatment groups or the placebo control group and monitored for a total of 24 weeks. Patients will return to the clinic each month for lab tests, and routine examinations.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤65 at study entry.
2. Is male, or female and, if female, meets all of the following criteria:

   1. Not breastfeeding
   2. Post-menopausal or negative serum pregnancy test result (human chorionic gonadotropin, beta subunit [β-hCG]) at Screening/Visit 1 (Day-7/Week-1) (not required for hysterectomized females)
   3. If of childbearing potential (including peri-menopausal women who have had a menstrual period within one year) must practice and be willing to continue to practice appropriate birth control (defined as a method which results in a low failure rate, i.e., less than 1% per year, when used consistently and correctly, such as double barrier methods [male condom with spermicide, with or without cervical cap or diaphragm], implants, injectables, oral contraceptives [must have been using for at least the last 3 months], some intrauterine contraceptive devices, tubal ligation, or in an established relationship with a vasectomized or same sex partner) during the entire duration of the study
3. Stable body weight (±5%) and health over the last 3 months.
4. Has a BMI between 30 kg/m2 and 45 kg/m2
5. Stable diet within the last three months
6. Subjects on antidepressants, excluding those listed in the exclusion criteria, must have been on a stable dose regiment for at least 3 months prior to study enrollment and maintain stable dose during the study
7. Clinical laboratory tests (hematology, clinical chemistry, and urinalysis) either normal, not clinically significant or with abnormalities consistent with obesity
8. Is able to read, understand, and sign the informed consent forms (ICF) and, when applicable, an authorization to use and disclose protected health information form (consistent with Health Insurance Portability and Accountability Act of 1996 [HIPAA] legislation), communicate with the investigator, and understand and comply with protocol requirements.

Exclusion Criteria:

1. Diagnosis of diabetes or on a diabetes medication
2. HbA1c ≥6.5% at Screening/Visit 1 (Day-7/Week-1)
3. Severe renal impairment (eGFR < 45 mg/mL/1.73 m2) and/or patients with acute or chronic metabolic acidosis. Acidosis is defined as >25mmol/L computed without K.

   Normal is 8- 16, but acidosis is >25
4. Use of any of the following medications in the eight weeks prior to entering screening for study participation and during the study:

   1. Use of any anti-diabetes medication including metformin and any combination drug that contains metformin
   2. Sildenafil
   3. Tadalafil
   4. Vardenafil
   5. OCT2/MATE inhibitors (e.g. cimetidine, quinidine, and pyrimethamine)
   6. Riociguat (guanylate cyclase stimulant)
   7. Alpha blockers
   8. Nitrates (e.g. oral nitrates, sublingual nitroglycerine and nitroglycerine patches)
   9. Potent CYP3A4 inhibitors (e.g. clarithromycin, telithromycin, nefazodone, itraconazole, ketoconazole, atazanavir, darunavir, indinavir, lopinavir, nelfinavir, ritonavir, saquinavir, tipranavir)
   10. All antihypertensive medications
   11. Medications associated with weight changes

       * Drugs approved for the treatment of obesity
       * Cypropheptadine or medroxyprogesterone
       * Atypical anti-psychotic drugs
       * Tricyclic antidepressants
       * Lithium, MAO's, glucocorticoids
       * SSRI's or SNRI's
       * Antiepileptic drugs
       * Systemic corticosteroids
       * Stimulants e.g. amphetamines
   12. Any dietary supplement that is labeled for weight management or maintenance of healthy weight
5. Diagnosis or evidence of eating disorders
6. ≥ 5% weight change in the last 3 months
7. Subjects who have had bariatric surgery
8. An infection requiring antibiotic treatment within the last 30 days
9. Any chronic inflammatory disease, e.g. inflammatory bowel disease rheumatoid arthritis, vasculitis, systemic lupus erythematosus
10. Diseases interfering with metabolism (including metabolism of branched chain amino acids) and/or ingestive behavior (myxedema, Cushing's disease, diabetes, schizophrenia, major psychoses, maple syrup urine disease, unmanaged depression etc.)
11. History of alcohol abuse (defined ≥ 21 drinks per week for males and > 14 drinks per week for females), within the past 3 months or failure on urinary drug screen
12. History of substance abuse (including alcohol abuse as defined above) in the past 12 months or a positive screen for drugs (opioids without a prescription), including marijuana, of abuse or alcohol at screening.
13. Has received any investigational drug within 3 months of Screening.
14. Has donated blood within 3 months before Screening or is planning to donate blood during the study (due to HbA1c reading at screening)
15. Other medical conditions that may diminish life expectancy to <2 years, including known cancers
16. Have been diagnosed with metastatic carcinomas in the last 5 years
17. Has known allergies or hypersensitivity to metformin, sildenafil or leucine
18. Have suffered myocardial infarction, stroke, arrhythmia in the last 6 months
19. Resting hypotension (BP <90/50 mmHg) or severe hypertension (BP >170/110 mmHg) If both or one of the parameters for diastolic or systolic BP is meet
20. Cardiac failure or coronary artery disease causing unstable angina
21. History or evidence at screening of left ventricular outflow obstruction (e.g., aortic stenosis, idiopathic hypertrophic subaortic stenosis) and those with severely impaired autonomic control of blood pressure
22. At risk for priapism due to anatomical deformation of the penis (e.g., angulation, cavernosal fibrosis, Peyronie's disease) or other conditions that predispose to priapism (e.g., sickle cell anemia, multiple myeloma, or leukemia)
23. Clinical evidence of hepatic impairment and/or ALT/AST >5X ULN
24. Is an immediate family member (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study at the clinical study site, or NuSirt Biopharma.
25. Is employed by NuSirt Biopharma (defined as an employee, temporary contract worker, or designee responsible for the conduct of the study).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Maximum of 70% female
Enrollment: 267 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2018-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zemel, PhD, Study Chair — NuSirt Biopharma
Locations (15):
- United States (15):
  - AMR, Mobile, Alabama
  - Catalina Research Institute, Montclair, California
  - Northern California Research, Sacramento, California
  - ACR, Meridian, Idaho
  - Synexus, Chicago, Illinois
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Clinical Trials Management, Metairie, Louisiana
  - Synexus, St Louis, Missouri
  - AMR, Las Vegas, Nevada
  - Rapid Medical Research, Cleveland, Ohio
  - Medical Research South, Charleston, South Carolina
  - Premier, Clarksville, Tennessee
  - Synexus, Dallas, Texas
  - Synexus, San Antonio, Texas
  - ACR, Jordan, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects meeting all inclusion criteria and no exclusion criteria were randomized to one of five treatment arms in the ratio of 1:1:1:1:1(A:B:C:D:E). The randomization was stratified by a maximum of 70% female with a BMI range between 30 kg/m2 and 45 kg/m2
Pre-assignment Details: The discrepancy in the number of enrolled subjects and the actual number that started the study is because some of the enrolled subjects did not start the study for the following reasons: they moved, were not compliant with investigator request or were sent on active military duty.
Groups:
- Leu Sil 1.0mg: 3 capsules BID consisting of 2 capsules containing 550 mg L-leucine each and 1 capsule containing 1.0 mg of sildenafil
  Leucine: 1100 mg BID
  Sildenafil Citrate 1.0 mg: Sildenafil 1.0 mg BID
- Leu Sil 4.0mg: 3 capsules BID consisting of 2 capsules containing 550 mg L-leucine each and 1 capsule containing 4.0 mg of sildenafil
  Leucine: 1100 mg BID
  Sildenafil Citrate 4.0 mg: Sildenafil 4.0 mg BID
- Leu Met Sil 1.0mg: 3 capsules BID consisting of 2 capsules containing 550 mg L-leucine and 250 mg metformin and 1 capsule containing 1.0 mg of sildenafil
  Leucine: 1100 mg BID
  Sildenafil Citrate 1.0 mg: Sildenafil 1.0 mg BID
  Metformin: Metformin 500 mg BID
- Leu Met Sil 4.0mg: 3 capsules BID consisting of 2 capsules containing 550 mg L-leucine and 250 mg metformin and 1 capsule containing 4.0 mg of sildenafil
  Leucine: 1100 mg BID
  Sildenafil Citrate 4.0 mg: Sildenafil 4.0 mg BID
  Metformin: Metformin 500 mg BID
Period: Overall Study
Arm/Group | Placebo | Leu Sil 1.0mg | Leu Sil 4.0mg | Leu Met Sil 1.0mg | Leu Met Sil 4.0mg
Started | 52 | 51 | 53 | 50 | 52
Completed | 42 | 40 | 42 | 37 | 41
Not Completed | 10 | 11 | 11 | 13 | 11
Not completed — Adverse Event | 3 | 4 | 1 | 2 | 0
Not completed — Lost to Follow-up | 7 | 7 | 10 | 11 | 11

BASELINE CHARACTERISTICS:
Population: Subjects who met the inclusion criteria, with BMI between 30kg/m2 and 45kg/m2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Leu Sil 1.0mg | Leu Sil 4.0mg | Leu Met Sil 1.0mg | Leu Met Sil 4.0mg | Total
Number analyzed (Participants) | 52 | 51 | 53 | 50 | 52 | 258
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 52 | 51 | 53 | 50 | 52 | 258
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.29 (11.30) | 40.94 (11.14) | 39.55 (11.14) | 41.36 (12.66) | 42.89 (10.70) | 41.20 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 29 | 32 | 39 | 35 | 173
  Male | 14 | 22 | 21 | 11 | 17 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 12 | 13 | 12 | 15 | 60
  Not Hispanic or Latino | 44 | 39 | 40 | 38 | 37 | 198
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 9 | 13 | 11 | 11 | 53
  White | 40 | 42 | 39 | 37 | 40 | 198
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 0 | 2
Weight (kg) [Mean (Standard Deviation); unit: kg] | 101.67 (13.856) | 105.05 (15.568) | 107.16 (17.962) | 100.18 (16.991) | 104.50 (17.405) | 103.74 (16.49)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 35.773 (3.31) | 37.179 (4.28) | 37.9 (4.20) | 36.425 (4.13) | 37.152 (4.23) | 36.89 (4.08)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 110.40 (10.998) | 112.91 (11.466) | 116.02 (12.411) | 111.17 (13.291) | 112.93 (13.311) | 112.71 (12.39)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Body Weight Change
Description: The percentage body weight change from baseline to Day 168 was evaluated.
Time Frame: Baseline to Day 168
Population: ANCOVA Analysis for Primary Endpoint - Percent Change in Body Weight from Baseline to Day 168 in per protocol population.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Placebo | Leu Sil 1.0mg | Leu Sil 4.0mg | Leu Met Sil 1.0mg | Leu Met Sil 4.0mg
Number analyzed (Participants) | 42 | 40 | 42 | 37 | 41
percentage | 1.121 (3.6241) | 0.674 (3.2286) | -0.489 (3.9041) | -0.929 (4.5533) | -0.552 (2.5924)
Statistical Analysis 1: Comparison: Placebo vs Leu Sil 1.0mg; Test type: Other — Analysis of covariance (ANCOVA) model: with treatment group and time as the main effects and baseline body weight as the covariate. Treatment A is used as the reference group; p = 0.5461, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Leu Sil 4.0mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0364, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Leu Met Sil 1.0mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0156, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs Leu Met Sil 4.0mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0349, ANCOVA

2. Secondary Outcome: Change in Absolute Body Weight
Description: The change in absolute body weight from baseline to day 168 was evaluated.
Time Frame: Baseline to Day 168
Population: ANCOVA Analysis for Secondary Endpoint - Change in Absolute Body Weight from Baseline to day 168 (Per-Protocol Population).
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | Leu Sil 1.0mg | Leu Sil 4.0mg | Leu Met Sil 1.0mg | Leu Met Sil 4.0mg
Number analyzed (Participants) | 42 | 40 | 42 | 37 | 41
kg | 1.126 (3.5903) | 0.678 (3.2502) | -0.460 (4.0352) | -0.870 (4.5445) | -0.461 (2.7583)
Statistical Analysis 1: Comparison: Placebo vs Leu Sil 1.0mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.5348, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Leu Sil 4.0mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0379, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Leu Met Sil 1.0mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0215, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs Leu Met Sil 4.0mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0464, ANCOVA

3. Secondary Outcome: Change in Percentage of Patients With ≥5% Body Weight Loss
Description: The number of patients with ≥5% body weight loss in each group was assessed from baseline to day 168.
Time Frame: Baseline to Day 168
Population: Analysis for Secondary Endpoint - Percentage of Subjects with ≥5% Relative Percentage Reduction from Baseline to day 168 in Body Weight by Treatment (Per-Protocol Population).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Leu Sil 1.0mg | Leu Sil 4.0mg | Leu Met Sil 1.0mg | Leu Met Sil 4.0mg
Number analyzed (Participants) | 42 | 40 | 42 | 37 | 41
Participants | 2 | 1 | 6 | 7 | 3
Statistical Analysis 1: Comparison: Placebo vs Leu Sil 1.0mg; Test type: Other — Pearson's Chi Square Test is used. Fisher exact test is used when any expected cell count is less than 5. Treatment A is used as the reference group; p = 1.0000, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs Leu Sil 4.0mg; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.2646, Chi-squared
Statistical Analysis 3: Comparison: Placebo vs Leu Met Sil 1.0mg; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.0749, Chi-squared
Statistical Analysis 4: Comparison: Placebo vs Leu Met Sil 4.0mg; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.6758, Chi-squared

4. Secondary Outcome: Change in Waist Circumference
Description: The change in waist circumference by using a tape measure across the mid-section was evaluated in subjects from baseline to day 168.
Time Frame: Baseline to Day 168
Population: ANCOVA Analysis for Secondary Endpoint - Change in Waist Circumference from Baseline (Per-Protocol Population).
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | Leu Sil 1.0mg | Leu Sil 4.0mg | Leu Met Sil 1.0mg | Leu Met Sil 4.0mg
Number analyzed (Participants) | 42 | 40 | 42 | 37 | 41
cm | 0.043 (5.5591) | 0.028 (5.5152) | -1.060 (5.5564) | -1.841 (4.7654) | 0.637 (5.7908)
Statistical Analysis 1: Comparison: Placebo vs Leu Sil 1.0mg; Test type: Other — Analysis of covariance (ANCOVA) model: with treatment group and time as the main effects and baseline waist circumference as the covariate. Treatment A is used as the reference group; p = 0.9656, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Leu Sil 4.0mg; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.4254, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Leu Met Sil 1.0mg; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.1276, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs Leu Met Sil 4.0mg; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.5937, ANCOVA

5. Secondary Outcome: Change in Total Cholesterol
Description: Changes in total cholesterol was examined by standard blood chemistry.
Time Frame: Baseline to Day 168
Population: ANCOVA Analysis for Secondary Endpoint - Change in Fasting Plasma Lipids from Baseline to day 168 (Per-Protocol Population).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Leu Sil 1.0mg | Leu Sil 4.0mg | Leu Met Sil 1.0mg | Leu Met Sil 4.0mg
Number analyzed (Participants) | 42 | 40 | 42 | 37 | 41
mg/dL | 1.0 (20.33) | 0.2 (20.96) | 1.9 (20.01) | -0.7 (16.74) | -6.6 (23.48)
Statistical Analysis 1: Comparison: Placebo vs Leu Sil 1.0mg; Test type: Other — Analysis of covariance (ANCOVA) model: with treatment group and time as the main effects and baseline fasting plasma lipid as the covariate. Treatment A is used as the reference group; p = 0.6010, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Leu Sil 4.0mg; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.6513, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Leu Met Sil 1.0mg; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.4354, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs Leu Met Sil 4.0mg; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.0310, ANCOVA

6. Secondary Outcome: Change in HDL Cholesterol
Description: Changes were measured in HDL cholesterol from Baseline to day 168 by standard blood chemistry.
Time Frame: Baseline, Day 168
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Leu Sil 1.0mg | Leu Sil 4.0mg | Leu Met Sil 1.0mg | Leu Met Sil 4.0mg
Number analyzed (Participants) | 42 | 40 | 42 | 37 | 41
mg/dL | 1.1 (7.43) | 0.6 (7.59) | 2.4 (6.40) | 1.8 (8.21) | 1.6 (7.72)
Statistical Analysis 1: Comparison: Placebo vs Leu Sil 1.0mg; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.4644, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Leu Sil 4.0mg; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.8573, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Leu Met Sil 1.0mg; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.8167, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs Leu Met Sil 4.0mg; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.9223, ANCOVA

7. Secondary Outcome: Change in LDL Cholesterol
Description: Changes in LDL Cholesterol was measured by standard blood chemistry from baseline to day 168.
Time Frame: Baseline, 168 days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Leu Sil 1.0mg | Leu Sil 4.0mg | Leu Met Sil 1.0mg | Leu Met Sil 4.0mg
Number analyzed (Participants) | 42 | 40 | 42 | 37 | 41
mg/dL | -5.5 (15.40) | -6.6 (16.86) | -4.2 (15.81) | -5.5 (11.77) | -11.6 (19.72)
Statistical Analysis 1: Comparison: Placebo vs Leu Sil 1.0mg; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.6574, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Leu Sil 4.0mg; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.8971, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Leu Met Sil 1.0mg; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.6317, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs Leu Met Sil 4.0mg; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.0341, ANCOVA

8. Secondary Outcome: Change in Triglycerides
Description: The change in triglycerides was evaluated by standard blood chemistry in subjects from Baseline to Day 168.
Time Frame: Baseline, Day 168
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Leu Sil 1.0mg | Leu Sil 4.0mg | Leu Met Sil 1.0mg | Leu Met Sil 4.0mg
Number analyzed (Participants) | 42 | 40 | 42 | 37 | 41
mg/dL | 13.4 (45.43) | 9.7 (56.42) | 1.9 (51.93) | -4.4 (47.02) | 3.5 (52.03)
Statistical Analysis 1: Comparison: Placebo vs Leu Sil 1.0mg; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.3720, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Leu Sil 4.0mg; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.2302, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Leu Met Sil 1.0mg; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.1377, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs Leu Met Sil 4.0mg; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.4295, ANCOVA

9. Secondary Outcome: Change in Plasma Glucose
Description: Change in plasma glucose was examined through standard fasting blood chemistry.
Time Frame: Baseline to Day 168
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Leu Sil 1.0mg | Leu Sil 4.0mg | Leu Met Sil 1.0mg | Leu Met Sil 4.0mg
Number analyzed (Participants) | 42 | 40 | 42 | 37 | 41
mg/dL | 0.4 (7.98) | -1.6 (9.35) | 0.3 (9.59) | 1.1 (12.43) | -1.7 (10.87)
Statistical Analysis 1: Comparison: Placebo vs Leu Sil 1.0mg; Test type: Other — Analysis of covariance (ANCOVA) model: with treatment group and time as the main effects and baseline Fasting Plasma Glucose as the covariate. Treatment A is used as the reference group; p = 0.6726, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Leu Sil 4.0mg; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.7934, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Leu Met Sil 1.0mg; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.5485, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs Leu Met Sil 4.0mg; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.3676, ANCOVA

10. Secondary Outcome: Change in Hemoglobin A1c (HbA1c)
Description: Change in Hemoglobin A1c was assessed in the subjects from baseline to day 168.
Time Frame: Baseline, Day 168
Population: ANCOVA Analysis for Secondary Endpoint - Change in HbA1c from Baseline to day 168 (Per-Protocol Population).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Placebo | Leu Sil 1.0mg | Leu Sil 4.0mg | Leu Met Sil 1.0mg | Leu Met Sil 4.0mg
Number analyzed (Participants) | 42 | 40 | 42 | 37 | 41
percentage of glycosylated hemoglobin | 0.16 (0.164) | 0.09 (0.167) | 0.11 (0.165) | 0.07 (0.198) | 0.09 (0.177)
Statistical Analysis 1: Comparison: Placebo vs Leu Sil 1.0mg; Test type: Other — Analysis of covariance (ANCOVA) model: with treatment group and time as the main effects and baseline HbA1c as the covariate. Treatment A is used as the reference group; p = 0.1653, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Leu Sil 4.0mg; Test type: Other — [test comment as in outcome 10, analysis 1]; p = 0.1970, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Leu Met Sil 1.0mg; Test type: Other — [test comment as in outcome 10, analysis 1]; p = 0.0608, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs Leu Met Sil 4.0mg; Test type: Other — [test comment as in outcome 10, analysis 1]; p = 0.1583, ANCOVA

11. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Diastolic blood pressure was measured by standard blood pressure monitor.
Time Frame: Baseline to Day 168
Population: ANCOVA Analysis for Secondary Endpoint - Change in Blood Pressure from Baseline to day 168 (Per-Protocol Population)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Leu Sil 1.0mg | Leu Sil 4.0mg | Leu Met Sil 1.0mg | Leu Met Sil 4.0mg
Number analyzed (Participants) | 42 | 40 | 42 | 37 | 41
mmHg | -1.7 (7.13) | 1.8 (9.57) | -2.6 (8.10) | 1.1 (9.16) | -3.3 (7.48)
Statistical Analysis 1: Comparison: Placebo vs Leu Sil 1.0mg; Test type: Other — Analysis of covariance (ANCOVA) model: with treatment group and time as the main effects and baseline diastolic blood pressure as the covariate. Treatment A is used as the reference group; p = 0.0524, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Leu Sil 4.0mg; Test type: Other — [test comment as in outcome 11, analysis 1]; p = 0.5221, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Leu Met Sil 1.0mg; Test type: Other — [test comment as in outcome 11, analysis 1]; p = 0.3702, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs Leu Met Sil 4.0mg; Test type: Other — [test comment as in outcome 11, analysis 1]; p = 0.5426, ANCOVA

12. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in Systolic blood pressure was assessed in patients from baseline to Day 168
Time Frame: Baseline, Day 168
Population: ANCOVA Analysis for Secondary Endpoint - Change in Blood Pressure from Baseline to day 168 (Per-Protocol Population).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Leu Sil 1.0mg | Leu Sil 4.0mg | Leu Met Sil 1.0mg | Leu Met Sil 4.0mg
Number analyzed (Participants) | 42 | 40 | 42 | 37 | 41
mmHg | -2.0 (9.97) | 0.5 (12.21) | -2.7 (9.12) | 0.6 (9.31) | -3.5 (9.29)
Statistical Analysis 1: Comparison: Placebo vs Leu Sil 1.0mg; Test type: Other — Analysis of covariance (ANCOVA) model: with treatment group and time as the main effects and baseline systolic blood pressure as the covariate. Treatment A is used as the reference group; p = 0.1843, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Leu Sil 4.0mg; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.4411, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Leu Met Sil 1.0mg; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.6991, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs Leu Met Sil 4.0mg; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.3721, ANCOVA

13. Secondary Outcome: Change in Inflammatory Markers
Description: hs-C-Reactive Protein (CRP) levels was examined by standard blood chemistry.
Time Frame: Baseline to Day 168
Population: Descriptive Statistics for Secondary Endpoint - hs-C-Reactive Protein Change from Baseline to day 168 (Per-Protocol Population).
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | Leu Sil 1.0mg | Leu Sil 4.0mg | Leu Met Sil 1.0mg | Leu Met Sil 4.0mg
Number analyzed (Participants) | 42 | 40 | 42 | 37 | 41
mg/L | 0.90 (2.401) | 0.12 (3.633) | 0.35 (3.385) | 0.56 (6.624) | 0.12 (3.551)
Statistical Analysis 1: Comparison: Placebo vs Leu Sil 1.0mg; Test type: Other — Analysis of covariance (ANCOVA) model: with treatment group and time as the main effects and baseline hsCRP as the covariate. Treatment A is used as the reference group; p = 0.0318, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Leu Sil 4.0mg; Test type: Other — [test comment as in outcome 13, analysis 1]; p = 0.3827, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Leu Met Sil 1.0mg; Test type: Other — [test comment as in outcome 13, analysis 1]; p = 0.0050, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs Leu Met Sil 4.0mg; Test type: Other — [test comment as in outcome 13, analysis 1]; p = 0.1045, ANCOVA

ADVERSE EVENTS:
Time Frame: 6 months
Description: Treatment-Emergent Adverse Event (TEAE) is defined as an adverse event occuring on (or) after the first dose of randomized Study medication, (or) existing prior to the time of and worsening after the time of the first dose of randomized study medication. N:number of subjects in the Intent-to-Treat population; n:number of subjects in the category; %:percentage calculated using the N as the denominator.
Arm/Group | Placebo | Leu Sil 1.0mg | Leu Sil 4.0mg | Leu Met Sil 1.0mg | Leu Met Sil 4.0mg
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/51 | 0/53 | 0/50 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 2/51 | 0/53 | 1/50 | 0/52
Other Adverse Events (participants affected / at risk) | 14/52 | 19/51 | 12/53 | 21/50 | 19/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=52) | Leu Sil 1.0mg (N=51) | Leu Sil 4.0mg (N=53) | Leu Met Sil 1.0mg (N=50) | Leu Met Sil 4.0mg (N=52)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=52) | Leu Sil 1.0mg (N=51) | Leu Sil 4.0mg (N=53) | Leu Met Sil 1.0mg (N=50) | Leu Met Sil 4.0mg (N=52)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
C-reactive protein increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Constipation (Renal and urinary disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Renal and urinary disorders) | 1 (1) | 2 (2) | 4 (4) | 21 (21) | 12 (12)
Headache (General disorders) | 4 (4) | 6 (6) | 0 (0) | 4 (4) | 5 (5)
Hypertension (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased Appetite (General disorders) | 2 (2) | 4 (4) | 2 (2) | 2 (2) | 3 (3)
Influenza (General disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Nausea (General disorders) | 1 (1) | 4 (4) | 1 (1) | 4 (4) | 6 (6)
Nasopharyngitis (General disorders) | 1 (1) | 5 (5) | 0 (0) | 1 (1) | 2 (2)
Pharyngitis (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6) | 2 (2) | 4 (4) | 4 (4)
Viral infection (General disorders) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT03364335/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT03364335/SAP_001.pdf